CLINICAL TRIAL: NCT07127081
Title: The Effect of Stress Ball and Watching Cartoons on Pain and Fear During Intravenous Catheter Application in Children: A Randomised Controlled Study
Brief Title: Intravenous Catheter Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Behire SANÇAR, Assist. Prof. Dr., Toros University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Toros University
Record Dates: First submitted 2025-08-04; First posted 2025-08-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: 6-12 Years Old
Keywords: Children; intravenous catheter; stress ball; cartoons; nursing

STUDY DESIGN:
Intervention Model Description: There will be tree groups (2 intervention, 1 control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stress ball (Experimental): Stress ball will be applied
  Interventions: Behavioral: Stress ball
- Cartoons (Experimental): Cartoons will be applied
  Interventions: Behavioral: Cartoons
- Control (No Intervention): No intervention will be made to this group.

INTERVENTIONS:
Behavioral: Stress ball — The study was a randomised controlled trial showing the effect of watching cartoons and squeezing a stress ball on pain and fear in children admitted for intravenous catheter insertion.
  Arms: Stress ball
Behavioral: Cartoons — The study was a randomised controlled trial showing the effect of watching cartoons and squeezing a stress ball on pain and fear in children admitted for intravenous catheter insertion.
  Arms: Cartoons

SUMMARY:
The study was a randomised controlled trial showing the effect of watching cartoons and squeezing a stress ball on pain and fear in children admitted for intravenous catheter insertion. Hypotheses of the Study Hypothesis 1: Children who watch cartoons during intravenous catheter insertion have lower pain and fear scores than the control group.

Hypothesis 2: The pain and fear of children who squeeze a stress ball during intravenous catheter insertion are lower than the control group Hypothesis 3: There is a difference between the pain and fear scores of children who watch cartoons and squeeze a stress ball.

DETAILED DESCRIPTION:
Explain how you determined the number The population of the study will consist of children admitted to the paediatric clinic of a State Hospital between 01 September 2025 and 01 February 2026. While calculating the sample size, the intergroup G*Power 3.1.9.4 maximum 10% type II error rate (1 - β = 0.90), maximum 5% type I error rate (α = 0.05), two-way hypothesis minimum sample size was determined as 90. It was planned to have 30 children in each group, with a total sample size of 90.

Implementation of Research:

Groups will be formed by computer-aided randomisation. Explanations will be made in accordance with the developmental level before the procedure. In the study, children will be divided into 3 groups as two intervention and one control group. The intervention groups are "Watching Cartoon Film" and "Squeezing Stress Ball". Cartoon Group: Two minutes before the intravenous catheter is inserted, the cartoon film chosen by the child will be started to be watched on the tablet. As a cartoon film, Puzzle Tower or Z Team on TRT Kids channel will be shown to children. Children will be able to watch the cartoon they want. The cartoons will be watched on a 10.2 inch iPad tablet provided by the researcher. Stress Ball Squeezing: Two minutes before the intravenous catheter is inserted, the stress ball will be squeezed. No intervention will be applied to the control group. Pain and fear scores of the child, parent and researcher will be recorded before, during and after the procedure. While the health professional performing the routine intravenous catheter procedure will intervene, the researcher will record the data before, during and after the procedure. The investigators will never perform the intravenous catheter insertion procedure. The researcher will collect relevant data from the child, parent and researcher during intravenous catheter insertion. The data will be recorded by Dr.Hem.Zühal Artuvan, one of the researchers. Consort Flow Diagram of the study is shown in Figure 1.

ELIGIBILITY:
Inclusion Criteria:

* Those who were admitted to Toros State Hospital, Child service on 01 September 2025- 01.02.2026,
* Children aged 6 to 12 years,
* Children scheduled for intravenous catheterisation,
* Children without mental and developmental retardation,
* Children who can speak and understand Turkish,
* Children and parents who signed an informed consent form.

Exclusion Criteria:

* Children who cannot speak or communicate in Turkish,
* Children whose first attempt to insert an intravenous catheter failed,
* Children and parents who did not sign the informed consent form.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Pain Scale | 22 weeks
  It is the most frequently used pain assessment method. Facial expressions are considered as reliable and unbiased markers. It was developed by Donna Wong and Connie Morain Baker in 1981 and revised in 1983. It is suitable to be applied at the age of three years and above. The pain level of the faces on the scale is explained to the child: "0= no pain.......10= unbearably severe pain". According to the scoring; 0-4 indicates mild pain, 5-6 indicates moderate pain, 7-8 indicates severe pain, 9-10 indicates unbearably severe pain. The administration time of the measurement tool is approximately 2 minutes [9,10,11].
Children's Fear Scale | 22 weeks
  It evaluates pain-related fear in children. The Child Fear Scale (CFS), developed by McMurty et al. (2011) and validated in Turkish by Özalp-Gerçeker et al. (2018), consists of five drawn facial expressions ranging from neutral expression (0=no anxiety) to frightened face (4=severe anxiety). In the validity-reliability study, the CQI value for the scale was found to be 0.89. The test-retest reliability (0.99) was found to be quite high. The scale cut-off point is 2 and scores of 2 and above are characterised as high level of fear. The Child Fear Scale is a valid and reliable measurement tool. The administration time of the measurement tool is approximately 2 minutes [12,13].

IPD SHARING:
Plan to Share IPD: No